CLINICAL TRIAL: NCT02799550
Title: Treatment of Elderly Relapsed and/or Refractory CD19-positive Acute Lymphoblastic Leukemia by Infusions of Allogeneic CART-19
Brief Title: Allogeneic CART-19 for Elderly Relapsed/Refractory CD19+ ALL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART-ALL-2015
Record Dates: First submitted 2016-05-31; First posted 2016-06-15 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2018-06

CONDITIONS: Leukemia
Keywords: CART; ALL; Relapsed; Refractory; CD19+
MeSH Terms: conditions — Leukemia; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- allogeneic CART-19 (Experimental): infusions of allogeneic CD19-directed chimeric antigen receptor-modified T cells (CART-19)
  Interventions: Biological: allogeneic CART-19

INTERVENTIONS:
Biological: allogeneic CART-19 — allogeneic CD19-directed chimeric antigen receptor-modified T cells (CART-19)

SUMMARY:
The purpose of this study is to evaluate the safety and efficiency of allogeneic cluster of differentiation 19 (CD19)-directed chimeric antigen receptor modified T cells (CART-19) infusions in patients with relapsed / refractory B-cell acute lymphoblastic leukemia (B-ALL)

DETAILED DESCRIPTION:
The relapsed and/or refractory B-ALL patients will receive infusions of allogeneic CART-19 within 1 week after chemotherapy. The re-induction chemotherapy regimen was primarily vindesine, mitoxantrone, cyclophosphamide, pegaspargase and dexamethasone, and no graft-versus-host disease (GVHD) prevention was conducted pre- and post- therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Patient with relapsed and/or refractory CD19 positive B-cell acute lymphoblastic leukemia (B-ALL)
* Estimated life expectancy ≥ 12 weeks (according to investigator's judgment)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2

Exclusion Criteria:

* Previous treatment with investigational gene or cell therapy medicine products
* CD19 negative B-cell leukemia
* Any uncontrolled active medical disorder that would preclude participation as outlined

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | 1 year
  defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment Adverse events assessed according to NCI-CTCAE v4.0 criteria

SECONDARY OUTCOMES:
Overall response rate of allogeneic CART-19 | up to 24 weeks
  An objective response is defined as: (1) a morphologic complete response (CR) or (2) a complete response with incomplete recovery of counts (CRi) (based on NCCN guidelines (National Comprehensive Cancer Network (NCCN), 2014) or (3) a negative minimal residual disease assessed by flow cytometry or qPCR
Disease-free survival | up to 24 weeks
Overall survival | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Huisheng Ai, MD, Study Chair — Affiliated Hospital of Academy of Military Medical Sciences
Locations (2):
- China (2):
  - Affiliated Hospital of Academy of Military Medical Sciences ,, Beijing, Beijing 100071
  - Chinese PLA General Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cai B, Guo M, Wang Y, Zhang Y, Yang J, Guo Y, Dai H, Yu C, Sun Q, Qiao J, Hu K, Zuo H, Dong Z, Zhang Z, Feng M, Li B, Sun Y, Liu T, Liu Z, Wang Y, Huang Y, Yao B, Han W, Ai H. Co-infusion of haplo-identical CD19-chimeric antigen receptor T cells and stem cells achieved full donor engraftment in refractory acute lymphoblastic leukemia. J Hematol Oncol. 2016 Nov 25;9(1):131. doi: 10.1186/s13045-016-0357-z. PMID 27887660